CLINICAL TRIAL: NCT06672276
Title: An Open, Parallel, Single-dose Phase I Clinical Study to Evaluate the Pharmacokinetics and Safety of TQD3606 for Injection in Subjects With Renal Insufficiency
Brief Title: To Evaluate the Pharmacokinetics and Safety of TQD3606 for Injection in Subjects With Renal Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQD3606-I-03
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Resistant to Gram-positive, Gram-negative and Anaerobic Bacteria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A: Subjects with mild renal insufficiency (Active Comparator): This group patients were given TQD3606 only one time
  Interventions: Drug: TQD3606
- B: Subjects with moderate renal insufficiency (Active Comparator): This group patients were given TQD3606 only one time
  Interventions: Drug: TQD3606
- C: Subjects with severe renal insufficiency (Active Comparator): This group patients were given TQD3606 only one time
  Interventions: Drug: TQD3606
- D: Health volunteers (Active Comparator): This group patients were given TQD3606 only one time
  Interventions: Drug: TQD3606

INTERVENTIONS:
Drug: TQD3606 — TQD3606 is a fixed-dose combination of meropenem and avibactam. Meropenem is a carbapenem antimicrobial agent, and avibactam is a β-lactamase inhibitor.

SUMMARY:
The study is an open, parallel, single-dose phase I clinical study to evaluate the pharmacokinetics and safety of TQD3606 for injection in subjects with renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet all of the following criteria for inclusion in this study:

* Understand the content, process and possible adverse reactions of the trial, be able to complete the study in accordance with the requirements of the trial protocol, and voluntarily sign the informed consent;
* Participants (including their partners) voluntarily used effective contraception within 3 months from 2 weeks before until the last use of study drug;
* Participants aged 18 ~ 75 ;
* Body mass index (BMI) and 18 or 32 kg/m2 or less, and the male weight 50 kg or greater, female weight 45 kg or more;

For renal impairment subjects, also required meet all of the following criteria for inclusion in this study:

* Subjects with moderate to severe renal insufficiency and end-stage renal disease were required to meet the diagnostic criteria for chronic kidney disease(CKD);
* Stable renal function: creatinine detection of at least two intervals of 3 days (30 days before the screening test results for the first time acceptable) inside and outside school or in our test result, and two detecting serum creatinine results before and after the fluctuation (calculation formula: (second results - 1)) / 1 time is less than 30%;
* During the screening period, the individual glomerular filtration rate (GFR, mL/min, using the modification of diet in renal disease( MDRD) formula, based on the results of the second serum creatinine test) was classified as follows: 60≤GFR≤89 mL/min (Group A, mild renal dysfunction, CKD2 period), or 30≤GFR≤59 mL/min (Group B, moderate renal dysfunction, CKD3 period), or 15≤GFR≤29 mL/min (Group C, severe renal dysfunction, CKD4 period).

Subjects in the normal renal function group must also meet the following criteria for inclusion in this study:

* Those who have normal results of laboratory examination, physical examination, 12-lead electrocardiogram (ECG), anterolateral chest x-ray and color ultrasound during the screening period, or those who are judged to be abnormal and non-clinically significant by the investigator;
* Individual glomerular filtration rate (GFR, mL/min, MDRD formula) during the screening period of subjects: GFR≥90 mL/min;

Exclusion Criteria:

All subjects were not eligible for the study if they met any of the following criteria:

* Those with allergies, or known history of allergy to meropenem or avibactam, known history of anaphylactic shock or other severe allergic reactions to penicillins, cephalosporins, carbapenems and other β-lactam antibiotics (such as epidermolysis bullosa atrophic dermatitis, exfoliative dermatitis), etc.;
* Those who have any type of treated or untreated malignant tumor (whether cured or not) within 5 years before screening or in the baseline period (except for basal cell carcinoma of the skin);
* Those who have serious digestive system, respiratory system, nervous system, blood system, endocrine system, tumor, immune, psychiatric or cardiovascular and cerebrovascular diseases within 1 year before screening, and are not suitable to participate in this trial as assessed by the investigator;
* Those who have major diseases or major surgeries within 4 weeks before dosing, or those who plan to undergo surgery during the study;
* Those who have donated (or lost blood) ≥ 400 mL within 3 months before screening, or have received blood products;
* Those who smoke more than 10 cigarettes per day on average in the 3 months before screening;
* History of substance abuse within 5 years prior to screening, and/or average weekly alcohol intake of more than 14 units (female subjects) or 21 units (male subjects) in the 3 months prior to screening (1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
* Those who have taken a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or excessive consumption of tea, coffee, grapefruit/grapefruit juice and/or caffeinated beverages (an average of more than 8 cups per day, each cup of 200 mL) within 2 weeks before dosing;
* Those who have ingested any products containing alcohol within 48 hours before receiving the study drug, or those who have a positive alcohol breath test;
* Drug abusers, or those who have used soft drugs (such as marijuana) within 3 months before screening, or who have taken hard drugs within 1 year before screening, or who have a positive urine drug screen at baseline;
* Active hepatitis B virus (HBV) () or hepatitis C virus (HCV) infection, or human immunodeficiency virus (HIV) antibody positive; or those who are positive for treponema pallidum antibodies ;
* Female subjects are lactating during the screening period or during the trial or have a positive serum pregnancy result;
* Other situations that the investigator considers unsuitable for enrollment.

Renal impairment subjects were not eligible for the study if they met any of the following criteria:

* Those who have participated in other clinical studies within 1 month before screening and have used any clinical investigation drugs or medical devices, the date of the last clinical study administration shall be used as the time benchmark (if it is a clinical investigation drug with a long half-life, at least 5 half-lives should be separated from the administration of this study);
* Patients with acute renal failure, with a history of kidney transplantation, or subjects who require kidney transplantation or undergo any type of dialysis during the expected trial;
* Obstructive urinary tract disease (e.g., urinary tract obstruction caused by urinary stones, urinary tract obstruction caused by abdominal mass lesions, etc.) or causes of renal impairment unrelated to renal parenchymal dysfunction (e.g., polycystic kidney, renal tumor, renal artery stenosis, drugs, severe infection, volume depletion, heart failure, etc.);
* People with urinary incontinence;
* At the time of screening, the therapeutic drugs and/or other treatment drugs for comorbidities have not met the requirements of stable medication for 1 month, or there are new drugs within 1 month (except for drugs used temporarily or intermittently, such as erythropoietin used once a month, or diuretics are temporarily required, etc.);
* Systolic blood pressure ≥ 160 mmHg or ≤80 mmHg, diastolic blood pressure ≥ 100 mmHg or ≤50 mmHg, and heart rate outside the range of 50-100 beats/minute (both ends inclusive) during the screening period or baseline period;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2× ULN (upper limit of normal, ULN) and total bilirubin > 1.5×ULN in the screening period or baseline period; albumin< 25 g/L; Absolute neutrophil value< 1.3×109/L; Hemoglobin < 80g/L; Platelet count< 80×109/L;
* Congestive heart failure with New York Heart Association(NYHA) grade III or IV, or left ventricular ejection fraction <50% at screening;

Normal subjects were excluded from the study if they met any of the following criteria:

* Those who have participated in other clinical studies within 3 months before screening and have used any clinical investigation drugs or medical devices, with the date of the last clinical study administration as the time benchmark (if it is a clinical investigation drug with a long half-life, there needs to be at least 5 half-lives between it and the administration of this study);
* Those who have used any drug within 14 days or 5 half-lives (whichever is longer) before dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  Peak blood drug concentration of meropenem and avibactam.
Area under the concentration-time curve (AUC) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  The area under the time curve of the plasma concentration -time curve of meropenem and avibactam.
Time-to-maximum concentration (Tmax) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  Time-to-maximum concentration of meropenem and avibactam.
Total body clearance (CLt) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  Total body clearance of meropenem and avibactam.
Renal clearance (CLr) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  Renal clearance of meropenem and avibactam.
Apparent volume of distribution (Vd/F) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  Volume of distribution based on the terminal phase of meropenem and avibactam.
Terminal elimination rate (λz) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  First-order rate constant associated with the terminal (log-linear) elimination phase of meropenem and avibactam.
Mean residence time (MRT) | Before administration, 0.5, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24 hours after administration
  The average time that the drug stays in the body of meropenem and avibactam.

SECONDARY OUTCOMES:
Amount Excreted in Urine as Unchanged Drug or Metabolite (Ae0-24) | 0h before administration and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48 hours after administration
  Ae0-24 of meropenem and avibactam.
Adverse event rate | Baseline up to 72 hours
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Qianfoshan Hospital), Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong